CLINICAL TRIAL: NCT04012632
Title: Polymorphisms in the Kisspeptin/GPR54 Pathway Genes and the Risk of Early Puberty
Brief Title: Kisspeptin/GPR54 Pathway and Early Puberty
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Di Li, Doctor, Shenzhen Center for Disease Control and Prevention
Other Study IDs: szCDC_1
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Puberty, Precocious
Keywords: SNP; kisspeptin; GPR54
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Early puberty cases of Han Chinese
- controls: Controls were matched to cases at 1:1 by age (± 3 months)
  Interventions: Other: this study was an observational study and no interventions were given to the participants

INTERVENTIONS:
Other: this study was an observational study and no interventions were given to the participants — the participants were recruited and the data as well as blood sample were collected.
  Groups: controls

SUMMARY:
There was a worldwide early trend in girls'age for puberty onset. The timing of puberty onset varies greatly among individuals, and much of this variation is modulated by genetic factors. This study was designed to explored the association of polymorphisms in KISS1/GPR54 pathway genes and the risk of early puberty in Chinese Han girls.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of central precocious puberty or early and fast puberty.

Exclusion Criteria:

* The participants who were not the first visit to the hospital and had been treated before.
* The participants who were with endocrine disorders.

Ages: 7 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Chinese Han girls from Shenzhen Children's Hospital or monitoring schools in Shenzhen
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
the polymorphism in the KISS1/GPR54 pathway genes | 3 months
  functional SNP loci of the KISS1/GPR54 pathway genes KISS1, KISSIR, PLCB1, PRKCA, and ITPR1 were selected and detected.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li D, Wu Y, Cheng J, Liu L, Li X, Chen D, Huang S, Wen Y, Ke Y, Yao Y, Su Z, Zhou L. Association of Polymorphisms in the Kisspeptin/GPR54 Pathway Genes With Risk of Early Puberty in Chinese Girls. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz229. doi: 10.1210/clinem/dgz229. PMID 32160304